CLINICAL TRIAL: NCT00317200
Title: Paclitaxel Plus Bevacizumab in Patients With Chemosensitive Relapsed Small Cell Lung Cancer (SCLC): A Safety, Feasibility and Efficacy Study
Brief Title: A Study of Paclitaxel Plus Bevacizumab in Patients With Chemosensitive Relapsed Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Genentech, Inc. (Industry); Walther Cancer Institute (Other)
Responsible Party: Nasser Hanna, M.D., Hoosier Oncology Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG LUN05-99
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator): Paclitaxel + Devacizumab in patients with chemosensitive relapsed small cell lung cancer.
  Interventions: Drug: Paclitaxel; Drug: Bevacizumab

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel 90 mg/m2 IV infusion over 1 hour, days 1, 8 and 15 of 28 day cycle.
Drug: Bevacizumab — Bevacizumab 10 mg/kg, days 1 and 15 of 28 day cycle

SUMMARY:
Improvements in therapy for relapsed SCLC are much needed. Paclitaxel has been previously tested and found to have significant single agent activity in relapsed SCLC, including in refractory patients. Angiogenesis plays an important role in SCLC, increased VEGF levels are associated with worse outcomes. Bevacizumab, a monoclonal antibody to VEGF, increase response rates and survival when combined with chemotherapy agents compared with the chemotherapy agent alone in NSCLC, breast cancer, and colorectal cancer. Paclitaxel plus bevacizumab, in the dose and schedule proposed in this study, improves response rates and progression free survival compared with paclitaxel alone in women with metastatic breast cancer. Therefore, we will be testing the safety, feasibility, and efficacy of this regimen in patients with chemosensitive relapsed SCLC.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

Paclitaxel 90 mg/m2 IV infusion over 1 hour days 1, 8 and 15 of 28 day cycle

Plus

Bevacizumab 10 mg/kg on days 1 and 15 of 28 day cycle.

* 1 cycle = 28 days (4 weeks)
* Disease assessments will be performed per RECIST every other cycle
* After a minimum of 4 cycles or a maximum of 6 cycles of combination chemotherapy, bevacizumab monotherapy may continue until disease progression or intolerable side effects

ECOG Performance Status 0 or 1

Hematopoietic:

* White blood cell count > 3,000 mm3
* Absolute neutrophil count (ANC) > 1,500 mm3
* Platelet count > 100,000 mm3
* International normalized ration (INR) of prothrombin time ≤ 1.2
* PTT no more than 5 seconds longer than the ULN

Hepatic:

* Bilirubin < 1.5 x ULN
* Aspartate aminotransferase (AST, SGOT) < 2.5 x ULN

Renal:

* Urine protein:creatinine ratio <1.0

Cardiovascular:

* No history of myocardial infarction or angina pectoris/anginal equivalent in the last 6 months. Note: The patient may be on anti-anginal medications if the symptoms have been entirely controlled for greater than 6 months.
* No history of uncontrolled congestive heart failure or uncontrolled hypertension

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic proof of small cell lung cancer
* Chemo-sensitive disease defined as relapsed after 60 days from completion of first line chemotherapy.
* Measurable disease according to RECIST and obtained by imaging within 28 days prior to being registered for protocol therapy.
* Must have received treatment with at least 1 but not more than 2 prior chemotherapy regimens. (At least one regimen must contain a platinum agent. Previous treatment with irinotecan is allowed.)
* Prior radiation therapy must be completed at least 21 days prior to being registered for protocol therapy, and toxicities due to radiation must have recovered to ≤ grade 1 or baseline prior to registration.
* Prior cancer treatment must be completed at least 21 days prior to being registered for protocol therapy and the subject must have recovered from the acute toxicity effects of the regimen prior to registration.

Exclusion Criteria:

* No treatment with any investigational agent within 30 days prior to being registered for protocol therapy.
* No history or radiographic evidence of CNS involvement by head CT or MRI within 42 days prior to registration.
* No history of seizures, transient ischemic attack or stroke.
* No clinically significant infections as judged by the treating investigator.
* No other active cancer except SCLC.
* No prior treatment with topoisomerase I inhibitor.
* No contraindications to the use of paclitaxel or bevacizumab as per the investigator's clinical judgment.
* Must not have grade 3 or greater peripheral neuropathy.
* Must not have had major surgical procedure, open biopsy, or significant traumatic injury within 28 days of being registered for protocol therapy.
* No anticipation of need for major surgical procedure during the course of the study.
* Patients may not have had a minor surgical procedure, placement of an access device or fine needle aspiration within 7 days prior to being registered for protocol therapy.
* No evidence of bleeding diathesis or coagulopathy.
* No history of deep vein thrombosis or pulmonary embolism.
* No full dose/therapeutic anticoagulation with either low molecular weight heparin or unfractionated heparin or coumadin within 10 days prior to registration.
* Patients must not have been using aspirin (>325 mg/day) or another nonsteroidal anti-inflammatory medications known to inhibit platelet function on a daily basis within 10 days prior to registration on study.
* Patients must not be using any of the following drugs known to inhibit platelet function within 10 days prior to registration: dipyridamole (Persantine), ticlopidine (Ticlid), clopidogrel (Plavix) and cilostazol (Pletal).
* Patients must not have a current non-healing wound or fracture.
* Patients must not have a history of or current hemoptysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To determine progression free survival(PFS) of this regimen in patients with chemosensitive relapsed small cell lung cancer (SCLC). | 18 months

SECONDARY OUTCOMES:
To determine the response rate of the combination of paclitaxel and bevacizumab with chemosensitive SCLC. | 18 months
To determine the toxicity of the combination of paclitaxel and bevacizumab in patients with SCLC. | 18 months
To determine overall survival. | 18 months
To assess VEGF polymorphisms in the study population. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, M.D., Study Chair — Hoosier Oncology Group, LLC
Locations (17):
- United States (17):
  - Highlands Oncology Group, Springdale, Arkansas
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Cancer Care Center of Southern Indiana, Bloomington, Indiana
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Center for Cancer Care at Goshen Health System, Goshen, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Quality Cancer Center (MCGOP), Indianapolis, Indiana
  - Community Regional Cancer Center, Indianapolis, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Center for Cancer Care, Inc., P.C., New Albany, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Siteman Cancer Center, St Louis, Missouri
  - Methodist Cancer Center, Omaha, Nebraska
  - Pennsylvania Oncology-Hematology Associates, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center Extramural Research Program, Rockledge, Pennsylvania

REFERENCES:
- [Result] Jalal S, Bedano P, Einhorn L, Bhatia S, Ansari R, Bechar N, Koneru K, Govindan R, Wu J, Yu M, Schneider B, Hanna N. Paclitaxel plus bevacizumab in patients with chemosensitive relapsed small cell lung cancer: a safety, feasibility, and efficacy study from the Hoosier Oncology Group. J Thorac Oncol. 2010 Dec;5(12):2008-11. doi: 10.1097/JTO.0b013e3181f77b6e. PMID 21102263
- See also: Hoosier Oncology Group Home Page — http://www.hoosieroncologygroup.org